CLINICAL TRIAL: NCT06179095
Title: The Effect of Virtual Reality on Anxiety During Intrauterine Device Insertion: Randomised Controlled Experimental Study
Brief Title: The Effect of Virtual Reality on Anxiety During Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Associate Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliED-4
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Intrauterine Device
Keywords: Virtual Reality; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental): Virtual reality to be applied to women undergoing intrauterine device insertion.
  Interventions: Other: Virtual reality
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practive on their own to reduce anxiety during intrauterine device insertion.

INTERVENTIONS:
Other: Virtual reality — Participants will view a specific relaxing and distracting scenario using virtual reality (VR) for approximately 7-8 minutes from one minute before the procedure until the end of the procedure. Assessment will be performed with STAI just before the intrauterine device insertion procedure, and again with STAI after the procedure.
  Arms: Virtual reality group

SUMMARY:
This study was planned to determine whether the use of virtual reality glasses during intrauterine device insertion has an effect on the anxiety level of women.

DETAILED DESCRIPTION:
Intrauterine device (IUD), which is one of the effective contraceptive methods in our country, is one of the known and frequently used methods. According to TDHS 2018 data, it was reported that 35% of women used IUD at some point in time, while the rate of women who were currently protected from pregnancy with IUD was 14% (TDHS, 2018). The fact that the rate of IUD use at any time is higher than the rate of current IUD users shows that the method is abandoned for various reasons (Kutlu & Kılıçaslan, 2014). However, although it is the most well-known method and used by one in three women in a period, the low rate of IUD use may be due to reasons such as the need to go to a health institution for application and controls, the feeling of embarrassment, discomfort and fear due to lack of information about the procedure, as well as known side effects (Kartal et al., 2013; Tan et al., 2022). However, in today's practice, no attempt is made to remove or reduce the discomfort of women, especially from vaginal examinations.

It is known that virtual reality glasses are used in many areas. The most frequently used of these is the health sector. It can be used for educational purposes as well as for treatment and rehabilitation purposes. It has been stated that with virtual reality applications in treatment and rehabilitation processes, patient motivation will increase and patient fear and anxiety will decrease (Holden, 2005; Riener & Harders, 2012;Öztürk & Sondaş, 2020).

In the light of the literature, it was determined that virtual reality goggles were not applied to reduce women's fear, anxiety and anxiety during IUD application. In this context, this study was planned to determine whether virtual reality goggles affect the anxiety level of women during IUD application.

ELIGIBILITY:
Inclusion Criteria:

* -Volunteering to participate in the research
* Answering questionnaire and scale forms completely
* Read and understand Turkish
* 18 years of age or older
* STAI score of 35 and above
* Not being pregnant,
* No complaints of acute pelvic pain,
* No damage or leysone in the perineum that may cause pain during examination,
* Not using a pharmacological agent or method with analgesic or anxiolytic effect 24 hours before the application,
* No vaginismus problem,
* Absence of a history of sexual abuse,
* Not having any physical or mental problems that may prevent communication.

Exclusion Criteria:

* -Not volunteering to participate in the research,
* Incomplete responses to questionnaires and scale forms
* Not understanding Turkish,
* Under 18 years of age
* Do not score less than 35 points on the STAI,
* Don't be pregnant,
* Complaint of acute pelvic pain,
* Any damage or leysone in the perineum that may cause pain during examination,
* Having used a pharmacological agent or method with analgesic or anxiolytic effect 24 hours before the application,
* Having a vaginismus problem,
* Previous history of sexual abuse,
* Having any physical or mental problem that prevents communication.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 80 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | between one to six months
  The form consists of questions about socio-demographic and intrauterine device insertion
The State/Trait Anxiety Inventory (STAI) | between one to six months
  This inventory was developed by Spielberg in 1973 and each of the subscales ranges from 1 (not at all) to 4 (very much). The lowest and highest scores that can be obtained from each subscale are 20 and 80, respectively. Higher scores are associated with more anxiety. The alpha value of the scale varies between 0.86 and 0.92 . Öner et al. 1983, it was shown that the alpha value of the Turkish version of the STAI ranged between 0.83 and 0.87.27.
Visual Anolag Scale (VAS) | between one to six months
  It was developed by Price et al. (1983) to assess the severity of pain (Price et al. 1983). It is a line, usually 10 cm long, horizontal or vertical, starting with "No Pain" and ending with "Intolerable Pain". This line may be just a straight line, or it may be divided into equal intervals, or it may have description words placed on the line to describe pain. It is generally accepted that the vertical line is easier to understand. The patient indicates the intensity of his/her pain with a mark on this line where he/she deems appropriate. The distance between the beginning of no pain and this point is measured in "cm" and recorded. Values vary between 0 and 10 and higher values indicate increased pain. Turkish validity and reliability was performed by Eti Aslan (Eti Aslan, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: remzire karadogan, Midwife, Principal Investigator — Kırklareli University
Locations (1):
- 1.Murat State Hospital, Edirne, Turkey (Türkiye)